CLINICAL TRIAL: NCT00057681
Title: Treatment of Early Age Mania (TEAM) Study
Brief Title: Study of Outcome and Safety of Lithium, Divalproex and Risperidone for Mania in Children and Adolescents
Acronym: TEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01MH064846-06 (NIH); U01MH064846 (NIH); U01MH064911 (NIH); U01MH064868 (NIH); U01MH064887 (NIH); U01MH064850 (NIH); U01MH064869 (NIH)
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Bipolar Disorder
Keywords: Mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Lithium Carbonate; Valproic Acid; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive treatment with lithium for 8 to 16 weeks
  Interventions: Drug: Lithium carbonate
- 2 (Experimental): Participants will receive treatment with valproate for 8 to 16 weeks
  Interventions: Drug: Valproate
- 3 (Experimental): Participants will receive treatment with risperidone for 8 to 16 weeks
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Lithium carbonate — Titrated until blood level is 1.1 to 1.3 mEq/L
  Arms: 1
Drug: Valproate — Titrated until blood level is 111 to 125 ug/mL
  Other Names: Depakote
  Arms: 2
Drug: Risperidone — Titrated by weight until dose is 2.0 mg BID to 3.0 mg BID
  Other Names: Risperdal
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness of the medications, lithium (Eskalith®), valproate (Depakote®), and risperidone (Risperdal®) in treating children and adolescents with bipolar disorder or symptoms of mania.

DETAILED DESCRIPTION:
Patients are randomly assigned to receive lithium (Eskalith), valproate (Depakote), or risperidone (Risperdal) for 8 to 16 weeks. They will have weekly visits to monitor their response to the medication. When the study is complete, care will be transferred to the child's treating psychiatrist.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for bipolar I (manic or mixed) or mania for at least 4 weeks
* CGAS less than or equal to 60
* Good physical health

Exclusion Criteria:

* Schizophrenia or any pervasive developmental disorder
* Major medical or neurological disease
* History of addiction to illicit substances or alcohol or drug abuse within the last 4 weeks
* IQ less than 70
* Pregnancy or breast-feeding
* Unacceptable methods of contraception
* In-patient care at baseline

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 379 (Actual)
Dates: Start 2003-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Geller, MD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pittsburgh/WPIC, Pittsburgh, Pennsylvania
  - University of Texas, Galveston, Texas

REFERENCES:
- [Background] Tillman R, Geller B, Klages T, Corrigan M, Bolhofner K, Zimerman B. Psychotic phenomena in 257 young children and adolescents with bipolar I disorder: delusions and hallucinations (benign and pathological). Bipolar Disord. 2008 Feb;10(1):45-55. doi: 10.1111/j.1399-5618.2008.00480.x. PMID 18199241
- [Result] Geller B, Luby JL, Joshi P, Wagner KD, Emslie G, Walkup JT, Axelson DA, Bolhofner K, Robb A, Wolf DV, Riddle MA, Birmaher B, Nusrat N, Ryan ND, Vitiello B, Tillman R, Lavori P. A randomized controlled trial of risperidone, lithium, or divalproex sodium for initial treatment of bipolar I disorder, manic or mixed phase, in children and adolescents. Arch Gen Psychiatry. 2012 May;69(5):515-28. doi: 10.1001/archgenpsychiatry.2011.1508. Epub 2012 Jan 2. PMID 22213771
- [Derived] Walkup JT, Wagner KD, Miller L, Yenokyan G, Luby JL, Joshi PT, Axelson DA, Robb A, Salpekar JA, Wolf D, Sanyal A, Birmaher B, Vitiello B, Riddle MA. Treatment of Early-Age Mania: Outcomes for Partial and Nonresponders to Initial Treatment. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):1008-19. doi: 10.1016/j.jaac.2015.09.015. Epub 2015 Oct 8. PMID 26598476
- [Derived] Salpekar JA, Joshi PT, Axelson DA, Reinblatt SP, Yenokyan G, Sanyal A, Walkup JT, Vitiello B, Luby JL, Wagner KD, Nusrat N, Riddle MA. Depression and Suicidality Outcomes in the Treatment of Early Age Mania Study. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):999-1007.e4. doi: 10.1016/j.jaac.2015.09.016. Epub 2015 Oct 8. PMID 26598475
- [Derived] Vitiello B, Riddle MA, Yenokyan G, Axelson DA, Wagner KD, Joshi P, Walkup JT, Luby J, Birmaher B, Ryan ND, Emslie G, Robb A, Tillman R. Treatment moderators and predictors of outcome in the Treatment of Early Age Mania (TEAM) study. J Am Acad Child Adolesc Psychiatry. 2012 Sep;51(9):867-78. doi: 10.1016/j.jaac.2012.07.001. Epub 2012 Jul 31. PMID 22917200
- [Derived] Tillman R, Geller B. Diagnostic characteristics of child bipolar I disorder: does the "Treatment of Early Age Mania (team)" sample generalize? J Clin Psychiatry. 2007 Feb;68(2):307-14. doi: 10.4088/jcp.v68n0218. PMID 17335331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from media advertisements and clinical referrals from 2003 to 2008. There were a total of N=379 subjects randomized to 1 of the 3 group strata. The strata were (1) medication-naive strategy, (2) add-on strategy, and (3) cross-taper strategy. Analyses have only been conducted on the N=279 subjects in the first stratum.
Groups:
- Randomized Medication - Lithium: Participants will receive treatment with lithium for 8 to 16 weeks. At the initial dispensing visit, dose was 150mg qHS for 2 days, then 150mg BID for subjects <25kg; 150mg BID for 2 days, then 300mg BID for subjects 25-50kg; 300mg BID for 2 days, then 300mg AM / 600mg PM for subjects >50kg. Dose was adjusted to achieve blood levels of 0.8 mEq/L at week 1, 0.9-1.0 mEq/L at weeks 2-3, and 1.1-1.3 mEq/L at weeks 4-7.
- Randomized Medication - Divalproex Sodium: Participants will receive treatment with divalproex sodium for 8 to 16 weeks. At the initial dispensing visit, dose was 125mg qHS for 2 days, then 125mg BID for subjects <25kg; 250mg qHS for 2 days, then 125mg AM / 250mg PM for subjects 25-50kg; 250mg qHS for 2 days, then 250mg BID for subjects >50kg. Dose was adjusted to achieve blood levels of 75 ug/ml at week 1, 100-110 ug/ml at weeks 2-3, and 111-125 ug/ml at weeks 4-7.
- Randomized Medication - Risperidone: Participants will receive treatment with risperidone for 8 to 16 weeks. At the initial dispensing visit, dose was 0.25mg qHS for 2 days, then 0.25mg BID for subjects <25kg; 0.25mg BID for 2 days, then 0.5mg BID for subjects 25-50kg; 0.25mg BID for 2 days, then 0.5mg BID for subjects >50kg. Dose was adjusted at weeks 2-3 to 0.5mg BID for subjects <25kg, 1.0mg BID for subjects 25-50kg and >50kg. Dose was adjusted at weeks 4-5 to 1.0mg BID for subjects <25kg, 1.5mg BID for subjects 25-50kg, 2.0kg BID for subjects >50kg. Dose was adjusted at weeks 6-7 to 2.0mg BID for subjects <25kg, 2.0mg AM / 3.0mg PM for subjects 25-50kg, 3.0mg BID for subjects >50kg.
Period: Overall Study
Arm/Group | Randomized Medication - Lithium | Randomized Medication - Divalproex Sodium | Randomized Medication - Risperidone
Started | 137 | 139 | 103
Completed | 72 | 67 | 69
Not Completed | 65 | 72 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Medication - Lithium | Randomized Medication - Divalproex Sodium | Randomized Medication - Risperidone | Total
Number analyzed (Participants) | 137 | 139 | 103 | 379
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 137 | 139 | 103 | 379
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.92 (2.79) | 9.85 (2.37) | 10.99 (2.95) | 10.19 (2.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 70 | 52 | 175
  Male | 84 | 69 | 51 | 204
Region of Enrollment [Number; unit: participants]
  United States | 137 | 139 | 103 | 379

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impressions-Bipolar Mania Improvement
Description: The Clinical Global Impressions-Bipolar (CGI-BP) assessment instrument measured improvement in mania, depression, and overall bipolar illness. The primary outcome measure was mania improvement, which measured the change in mania from baseline. Scores were 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: Measured at Week 8
Population: CGI-BP mania improvement data were analyzed for all subjects completing 8 weeks of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Medication - Lithium | Randomized Medication - Divalproex Sodium | Randomized Medication - Risperidone
Number analyzed (Participants) | 72 | 67 | 69
units on a scale | 2.49 (1.05) | 2.73 (1.08) | 1.70 (0.63)

2. Secondary Outcome: Modified Side Effects Form for Children and Adolescents
Description: The Modified Side Effects Form for Children and Adolescents includes 62 potential side effects, with measures of frequency and severity for each item. Frequencies are 0=not present, 1=1-2 days, 2=3-4 days, 3=5-7 days. Severity scores are 0=not present, 1=mild (does not interfere with functioning), 2=moderate (some interference with functioning), 3=severe (functioning is significantly impaired because of side effects). Items for cardiovascular, gastrointestinal, central nervous system, ocular, mouth and nose, genito urinary, dermatology, musculo-skeletal, and other side effects are included. For analyses, side effects that were reported at any frequency and a severity of 2 or greater were considered present.
Time Frame: Measured at Week 8
Population: Modified Side Effects Form for Children and Adolescents data were analyzed for all subjects completing 8 weeks of the study.
Measure: Mean (Standard Deviation); unit: side effects at week 8
Arm/Group | Randomized Medication - Lithium | Randomized Medication - Divalproex Sodium | Randomized Medication - Risperidone
Number analyzed (Participants) | 72 | 67 | 69
side effects at week 8 | 5.11 (3.54) | 4.95 (3.29) | 3.70 (2.42)

3. Secondary Outcome: K-SADS Mania Rating Scale
Description: The K-SADS Mania Rating Scale (KMRS) is comprised of 15 items modified from WASH-U-KSADS items. The individual items are scored on a 1-6 severity scale and then these item scores are summed to create an overall KMRS score. Guidelines for interpretation are as follows: 0-11 = no or minimal mania, 12-17 = mild mania, 18-25 = moderate mania, 26+ = marked or worse mania. The maximum possible score is 64.
Time Frame: Measured at Week 8
Population: KMRS data were analyzed for all subjects completing 8 weeks of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Medication - Lithium | Randomized Medication - Divalproex Sodium | Randomized Medication - Risperidone
Number analyzed (Participants) | 72 | 67 | 69
units on a scale | 24.06 (12.11) | 26.31 (11.71) | 14.58 (7.47)

ADVERSE EVENTS:
Arm/Group | Randomized Medication - Lithium | Randomized Medication - Divalproex Sodium | Randomized Medication - Risperidone
Serious Adverse Events (participants affected / at risk) | 6/137 | 4/139 | 5/103
Other Adverse Events (participants affected / at risk) | 0/137 | 0/139 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Medication - Lithium (N=137) | Randomized Medication - Divalproex Sodium (N=139) | Randomized Medication - Risperidone (N=103)
Hospitalization (Psychiatric disorders) | 5 (5) | 4 (4) | 5 (5) — Admission to the hospital or prolongation of a hospital stay results because of the adverse event.
Event requiring intervention to prevent permanent impairment or damage (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — A condition that requires medical or surgical intervention to preclude permanent impairment or damage to a subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No